CLINICAL TRIAL: NCT01361529
Title: Phase 1 Study of FLP Injection on Tumor Patients
Brief Title: Safety Study of FLP Injection to Treat Tumor Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acea Bio (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Wanhong Xu,Deputy General Manager, Acea Bio (Hangzhou) Co., Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACEA100108(FLP)
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Advanced Cancer
Keywords: dose escalation
MeSH Terms: interventions — fluorapacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- safty test (Experimental): FLP,dose escalation,MTD
  Interventions: Drug: FLP,dose escalation,MTD

INTERVENTIONS:
Drug: FLP,dose escalation,MTD — dosage from 93mg/m2 to 331mg/m2, 7 days' continuous dosing, 21 days for one cycle
  Other Names: Fluorapacin

SUMMARY:
The purpose of this study is to determine the tolerance and maximum tolerated dose (MTD) for FLP Injection with multiple dose in tumor patients.

DETAILED DESCRIPTION:
To determine the tolerance and MTD for FLP Injection with multiple dose in tumor patients.

To test clinical pharmacokinetics (PK) and PK parameter

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 70 years old, male or female;
* histologically or cytologically proven advanced malignant solid tumors;
* cancer patients after conventional treatment failure and lack of effective treatment, or patients refusing effective treatment of existing practices;
* patients receiving the last treatment (chemotherapy, radiotherapy, biological therapy, targeted therapy, or other study drugs) for at least 4 weeks;
* expected survival time>3 months;
* ECOG score 0-1

Exclusion Criteria:

* viral activity in patients
* allergic to drugs or excipients;
* hypersensitivity to paclitaxel injection patients;
* HIV antibody positive, or suffering from other acquired and congenital immune deficiency disease, or history of organ transplantation;
* neutrophil count <1.5 × 109 / L, platelets <100 × 109 / L, or hemoglobin <90g / L;
* normal serum creatinine higher than 1.5 times the upper limit of reference range or the muscle of liver clearance <60ml/min;
* no case of liver ALT or AST> 2.5 times the upper limit of normal, or liver metastases than normal under the ALT or AST 5 times upper limit of reference range;
* fever or body temperature above 38 ℃ can be clinically significant impact on clinical trials of active infection;
* medications failed to control hypertension (systolic pressure is over 160 mmHg or diastolic pressure over 100mmHg);
* significant cardiovascular abnormalities (such as myocardial infarction, superior vena cava syndrome), or clinically significant arrhythmias (such as long QT syndrome, Corrected QTc not be measured or ≧ 480 ms);
* calcium, potassium, magnesium ions below the lower limit of normal;
* > I-level peripheral neuropathy
* Prior to the toxicity of anticancer therapy has not been restored or not from the surgery before full recovery;
* bone metastases for the primary lesion of palliative radiotherapy;
* any clinical problems can not control (such as the serious mental, neurological, cardiovascular, respiratory and other diseases);
* a tumor metastasis, or a variety of mental disorders center; no history of asthma;
* pregnancy or breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
adverse effect assessment | 21 days
  to evlauate the symptom of adverse effect and the number of participates with adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: jianying zhou, professor, Principal Investigator — First Affiliated Hospital of Zhejiang University; nong xu, professor, Principal Investigator — First Affiliated Hospital of Zhejiang University; jianzhong shentu, professor, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- GCP center,First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China